CLINICAL TRIAL: NCT03825952
Title: Optimizing mHealth for Adherence Monitoring and Intervention
Acronym: OAsIS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Jessica Haberer, MD, Director of Research, Massachusetts General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: K24MH114732 (NIH)
Record Dates: First submitted 2019-01-30; First posted 2019-02-01 (Actual); Last update posted 2022-12-12 (Actual); Status verified 2022-12

CONDITIONS: HIV/AIDS
Keywords: adherence
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Participants using MERM device (Experimental): Participants will use an electronic medication monitor to measure their adherence to ART in routine clinical care.
  Interventions: Device: MERM - medication event reminder monitor

INTERVENTIONS:
Device: MERM - medication event reminder monitor — The MERM will help measure adherence to ART in routine clinical care.

SUMMARY:
High and sustained adherence is critical for achieving the individual and public health benefits of HIV antiretroviral therapy (ART). Electronic adherence monitors provide a detailed understanding of adherence and enable real-time interventions. Research has shown the benefit of these monitors and low-cost models have recently become available; however, their use to date has largely been confined to the research context.

This study is an implementation science-driven assessment of strategies to improve uptake of electronic adherence monitoring and associated interventions for routine, clinical delivery of ART in Uganda. The study consists of two aims. In Aim 1, the investigators will conduct multi-level formative interviews to design a preliminary implementation strategy. In Aim 2, the investigators will use an iterative approach to optimize the implementation strategy. All work will be guided by the Consolidated Framework for Research Implementation.

DETAILED DESCRIPTION:
Design: Prospective mixed-method assessment with iterative improvements for program implementation

Populations: 1) Health care administrators and clinicians and 2) individuals taking ART

Study site: Kabwohe Clinical Research Centre (KCRC)

Approach The electronic adherence monitors to be assessed in this study are pill containers that record each opening as a proxy for pill taking behavior. They provide day-to-day information about adherence that can be used to provide informed counseling at clinic visits, as well as SMS reminders and notifications for missed or late doses. For Aim 1, the study team will recruit up to 35 health care administrators and clinicians from various levels of the Ugandan health care system (Health Center IV to the national hospital level), as well as 15 individuals taking ART at the KCRC. Research assistants will conduct individual, in depth qualitative interviews to define a preliminary implementation strategy for these electronic adherence monitors to be used in routine HIV clinical care. In Aim 2 (iteration 1), investigators will deploy the electronic adherence monitors and associated interventions per the strategy identified in Aim 1 among 30 individuals taking ART at the KCRC. Study staff will monitor their adherence for 3 months, during which time they will quantify multiple metrics of the deployment. The investigators will review these metrics with the same health care administrators and clinicians from Aim 1, as well as up to 15 individuals who used the adherence monitors in the Aim 2 deployment. Research assistants will then interview both groups to develop an improved implementation strategy for deployment in a second iteration. In Aim 2 (iteration 2), study staff will utilize the revised implementation strategy to deploy the electronic adherence monitors and associated interventions among a new cohort of 30 individuals taking ART at the KCRC. The study team will then repeat the assessment of the implementation strategy with the same health care administrators and clinicians from Aims 1 and 2 (iteration 1), as well as up to 15 individuals who used the adherence monitors in the Aim 2 (iteration 2) deployment. The investigators will conclude the study with recommendations for wide-scale uptake of this technology in routine HIV clinical care.

Aims Aim 1. Define a preliminary implementation strategy for real-time electronic adherence monitoring plus associated interventions for routine HIV clinical care in Uganda

Aim 2. Deploy and optimize an implementation strategy for real-time electronic ART adherence monitoring plus associated interventions in routine HIV clinical care in Uganda

ELIGIBILITY:
Inclusion Criteria:

* age >18 years
* engagement in HIV care
* For individuals taking ART:
* HIV infection per clinic records
* own a cellular phone

Exclusion Criteria:

* unwillingness or inability to provide informed consent
* intention to move >100 km away from KCRC during the three-month study period

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 174 (Actual)
Dates: Start 2018-03-28 (Actual); Primary Completion 2022-08-05 (Actual); Study Completion 2022-08-05 (Actual)

PRIMARY OUTCOMES:
Adherence to ART | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Jessica Haberer, MD, MS, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Kabwohe Clinical Research Center, Kabwohe, Sheema District, Uganda

REFERENCES:
- [Derived] Adong J, Asiimwe S, Nansera D, Muyindike W, Tumuhairwe JB, Baijuka R, Tindimwebwa E, Garrison LE, Haberer JE. Electronic Antiretroviral Therapy Adherence Monitors and Associated Interventions Improve Adolescent-Caregiver Relationships and Self-Efficacy Among Adolescents and Young Adults with HIV in Uganda. AIDS Patient Care STDS. 2023 Oct;37(10):489-494. doi: 10.1089/apc.2023.0164. PMID 37862075
- [Derived] Haberer JE, Baijuka R, Tumuhairwe JB, Tindimwebwa EB, Tinkamanyire J, Tuhanamagyezi E, Musoke L, Garrison LE, DelSignore M, Musinguzi N, Asiimwe S. Implementation of Electronic Adherence Monitors and Associated Interventions for Routine HIV Antiretroviral Therapy in Uganda: Promising Findings. Front Digit Health. 2022 Jul 22;4:899643. doi: 10.3389/fdgth.2022.899643. eCollection 2022. PMID 35937420
- [Derived] Haberer JE, Garrison L, Tumuhairwe JB, Baijuka R, Tindimwebwa E, Tinkamanyire J, Burns BF, Asiimwe S. Factors Affecting the Implementation of Electronic Antiretroviral Therapy Adherence Monitoring and Associated Interventions for Routine HIV Care in Uganda: Qualitative Study. J Med Internet Res. 2020 Sep 10;22(9):e18038. doi: 10.2196/18038. PMID 32687473